CLINICAL TRIAL: NCT02552563
Title: Engaging Caregivers in the Care of Veterans With Dementia
Brief Title: Engaging Caregivers in Dementia Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shahrzad Mavandadi, Research Health Science Specialist, Corporal Michael J. Crescenz VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01247
Record Dates: First submitted 2015-09-04; First posted 2015-09-17 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Standard care received by veterans in the Corporal Michael J. Crescenz VA Medical Center
- Dementia Care Management (Active Comparator): CG education, continuous support, communication and coping skills training, and veteran monitoring, via CG report, of medication, symptoms, and service needs.
  Interventions: Behavioral: Dementia Care Management

INTERVENTIONS:
Behavioral: Dementia Care Management — The intervention involves two main components. The first component includes individualized dementia care management that involves regular and extended contact between the CG, care manager, and when appropriate, Veteran's primary care provider (PCP). The care manager monitors Veterans' symptoms via CG report, provides psychoeducation and support to CGs, influences adherence to guidelines by providing timely and tailored information to PCPs, and suggests appropriate care strategies and service referrals. The second major component is the Telehealth Education Program (TEP). For this pilot study, the program was modified for use with individual CGs and was formatted so that CGs could select from a menu of up to 7 modules covering various content areas evaluated during the course of the care management assessments (e.g., communication skills, behavioral management techniques, stress management and coping skills, long-term planning, etc.).
  Other Names: Telehealth Education Program
  Arms: Dementia Care Management

SUMMARY:
This pilot study seeks to examine the extent to which, relative to usual care, a dementia care management program for veterans and their caregivers (CGs)improves patient (e.g., behavioral symptoms, delayed nursing home placement) and caregiver (e.g., CG mastery, burden, affect) outcomes.

DETAILED DESCRIPTION:
Dementia care guidelines and pharmacological and non-pharmacological treatments have been shown to reduce symptom burden and rates of institutionalization for individuals with dementia. However, there remain a variety of factors that complicate dementia care management in primary care settings. Patient-centered, integrated care management programs that involve caregiver (CG) education and psychosocial support may help facilitate access to and use of services and improve outcomes. The aims of this pilot were to examine 1) whether, relative to usual care (UC), a dementia care management program is associated with improved CG (e.g., mastery, burden, affect) and patient (e.g., behavioral symptoms) outcomes, 2) if, relative to UC, participants enrolled in the program have greater perceived access to and use of medical, social, and community/VA services, and 3) whether the dementia care management program is feasible and acceptable to participants.

ELIGIBILITY:
Inclusion Criteria:

* Patient and caregiver 18 years of age or older
* Patient is community dwelling
* Patient has a confirmed dementia diagnosis and/or significant cognitive impairment (per provider or CG report) that is verified upon the RA's cognitive screening assessment (per veteran (BOMC, score of 16 or above) or informant (AD8, score of 2 or above) and/or chart review
* CG lives with and/or provides care for the patient for an average of at least 4 hours per day.
* Veteran provides assent to contact his/her representative to pursue study participation
* Veteran representative as caregiver is willing and able to provide informed consent

Exclusion Criteria:

* Cognitive, hearing, visual, or other physical impairments leading to difficulty with assent/ informed consent process and/or assessment (veteran or caregiver)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Revised Memory and Behavior Problems Checklist (RMBPC) | Change in frequency and distress from baseline to 3 and 6 month follow-up
  Frequency of care recipient dementia-related behaviors and associated caregiver distress
Neuropsychiatric Inventory Questionnaire (NPI-Q) | Change in frequency and distress from baseline to 3 and 6 month follow-up
  Frequency of care recipient neuropsychiatric symptoms and associated caregiver distress
Zarit Burden Interview | Change in burden from baseline to 3 and 6 month follow-up
  Perceived caregiver burden

SECONDARY OUTCOMES:
Pearlin Stress and Coping Scale | Change in coping skills from baseline to 3 and 6 month follow-up
  Caregiver coping strategies
Lawton Caregiving and Stress Process Scales | Change in caregiver mastery from baseine to 3 and 6 month follow-up
  Caregiver mastery

CONTACTS AND LOCATIONS:
Overall Officials: Shahrzad Mavandadi, PhD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center
Locations (1):
- Philadelphia VA Medical Center, Philadelphia, Pennsylvania, United States